CLINICAL TRIAL: NCT03742141
Title: Intraoperative Video Laryngoscopy as Adjunct for Nerve Monitoring
Acronym: IOVL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: NeuroVision (Industry)
Responsible Party: Principal Investigator, Randall Owen, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: GCO 17-2617
Record Dates: First submitted 2018-11-12; First posted 2018-11-15 (Actual); Results first posted 2023-10-02 (Actual); Last update posted 2023-10-02 (Actual); Status verified 2023-08

CONDITIONS: Vocal Cord Function in Neck Procedures
Keywords: Thyroidectomy; Neck Procedures; Nerve Monitoring
MeSH Terms: interventions — Glycopyrrolate

STUDY DESIGN:
Intervention Model Description: All patients enrolled in the study will be in a single group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Intraoperative Video Laryngoscopy (Experimental): Participants undergoing neck procedures
  Interventions: Device: Intraoperative Video Laryngoscopy; Drug: Glycopyrrolate

INTERVENTIONS:
Device: Intraoperative Video Laryngoscopy — The IOVL is a disposable, otherwise standard fiberoptic laryngoscope that is inserted alongside the endotracheal tube following intubation for surgical procedures.
  Other Names: IOVL
Drug: Glycopyrrolate — 0.004mg/kg as per routine prior to intubation

SUMMARY:
The purpose of this study is to describe the impact of adding intraoperative video laryngoscopy (IOVL) to intraoperative laryngeal nerve monitoring (IOLNM) during neck procedures when IOLNM is routinely used, including thyroidectomy and re-operative parathyroidectomy. Specifically, the study team seeks to assess how frequently the use of IOVL provided confirmatory or additional information that may affect surgeon decision-making when IOLNM alone is ambiguous, or when there is equipment malfunction or failure. The IOVL is a disposable, otherwise standard fiberoptic laryngoscope (Larynxview, Neurovision Medical, Ventura CA) that is inserted alongside the endotracheal tube following intubation for surgical procedures. It allows assessment of vocal cord movement in response to nerve stimulation. Currently, the use of IOLNM is based on audio cues, and visual assessment of external laryngeal muscle movement during surgery in response to stimulation, but no direct assessment of vocal cord movement is routinely possible. This information can be ambiguous and subject to judgement of the surgeon. The addition of IOVL provides direct assessment to vocal cord movement in response to stimulus, and may be useful in light of ambiguous IOLNM data, or limited visualization of external laryngeal muscles.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older with capacity to make all medical decisions
* Medical indication for partial or total thyroidectomy, re-operative parathyroidectomy, or neck dissection

Exclusion Criteria:

* Patients who are under the age of 18
* Patients who are not able to make medical decisions or consent to research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2018-10-17 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall Owen, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (5):
- United States (5):
  - Mount Sinai Queens, Long Island City, New York
  - Mount Sinai Beth Israel, New York, New York
  - Mount Sinai West, New York, New York
  - Mount Sinai St. Luke's, New York, New York
  - The Mount Sinai Hospital, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intraoperative Video Laryngoscopy
Started | 125
Completed | 75
Not Completed | 50
Not completed — no surgery or post-operative laryngoscopy | 50

BASELINE CHARACTERISTICS:
Arm/Group | Intraoperative Video Laryngoscopy
Number analyzed (Participants) | 75
Age, Continuous [Mean (Full Range); unit: years] | 52.1 [23 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 52
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 20
  More than one race | 19
  Unknown or Not Reported | 18
BMI [Mean (Full Range); unit: kg/m^2] | 28.7 [18.5 to 46.3]
History of Thyroiditis [Count of Participants; unit: Participants] | 13
Thyroid Weight [Mean (Full Range); unit: grams] | 28.0 [2 to 200]
Thyroid Size [Mean (Full Range); unit: cm] | 5.4 [2 to 12.9]
Indication for surgery [Count of Participants; unit: Participants]
  Cancer | 21
  Nontoxic Multinodular Goiter | 15
  Toxic Multinodular Goiter | 3
  Suspicious Nodule | 14
  Grave's Disease | 4
  Other | 18
Type of surgery [Count of Participants; unit: Participants]
  Right hemithyroidectomy | 24
  Left hemithyroidectomy | 18
  Total thyroidectomy | 33

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Congruence of Nerve Integrity and Vocal Cord Functions
Description: Frequency of congruence - IOVL used in conjunction with routine intraoperative nerve monitoring to provide additional data on nerve integrity and vocal cord functions for patients undergoing neck procedures that place the recurrent and superior laryngeal nerves at risk for injury or postoperative dysfunction.
  Video-captured vocal cord movement as well as the Nerveana Power Index (NPI) audio signal were recorded. Loss of signal was considered any NPI value <100, which corresponds to loss of audio signal. The NPI is specific to the Nerveana machine, and is an index of the nerve/muscle response power (or area under the curve) as a percentage of the threshold level of response. Thus, positive EMG signal (EMG+) was an NPI value >100. Positive IOVL (IOVL+) correlated with observed vocal cord movement on nerve stimulation; negative IOVL indicated no visible vocal cord movement. Discordances were considered to be contradictory IOVL and EMG (e.g., IOVL+ EMG-) findings for a particular nerve.
Time Frame: up to 3 months post-resection
Measure: Count of Units; unit: nerves at risk
Units Other Than Participants: nerves at risk
Groups:
- Intraoperative Video Laryngoscopy: 75 participants (108 nerves at risk) undergoing thyroid lobectomy or total thyroidectomy for benign and malignant disease with concurrent use of intraoperative video laryngeal monitoring and intermittent standard EMG monitoring, using the Nerveana nerve monitoring system.
Arm/Group | Intraoperative Video Laryngoscopy
Number analyzed (Participants) | 75
Number analyzed (nerves at risk) | 108
nerves at risk
  EMG+ IOVL+ | 68
  EMG+ IOVL- | 13
  EMG- IOVL- | 17
  EMG- IOVL+ | 10

ADVERSE EVENTS:
Time Frame: 3 months
Description: Definition of adverse event from 21 CFR 312.32 (a): any untoward medical occurrence associated with the use of an intervention in humans, whether or not considered intervention-related.
Arm/Group | Intraoperative Video Laryngoscopy
All-Cause Mortality (participants affected / at risk) | 0/75
Serious Adverse Events (participants affected / at risk) | 1/75
Other Adverse Events (participants affected / at risk) | 2/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intraoperative Video Laryngoscopy (N=75)
Tracheostomy (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Intraoperative Video Laryngoscopy (N=75)
Transected nerve intraoperatively (Injury, poisoning and procedural complications) | 1
reintubation and a tracheostomy immediately postoperatively (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2022-01-18): https://cdn.clinicaltrials.gov/large-docs/41/NCT03742141/Prot_001.pdf